CLINICAL TRIAL: NCT03665597
Title: A Phase 1 Randomized Clinical Study of Pembrolizumab (MK-3475) to Evaluate the Relative Bioavailability of Subcutaneous Injection Versus Intravenous Infusion in Participants With Advanced Melanoma (KEYNOTE-555)
Brief Title: Relative Bioavailability Study of Subcutaneous Injection Versus Intravenous Infusion of Pembrolizumab (MK-3475) in Participants With Advanced Melanoma (MK-3475-555/KEYNOTE-555)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3475-555; MK-3475-555 (Other: MSD); KEYNOTE-555 (Other: MSD); 2019-001052-19 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-09-11 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Programmed Cell Death 1; PD1; PD-1; Programmed Cell Death-Ligand 1; PDL1; PD-L1
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort A Pembrolizumab Treatment Sequence 1 (Experimental): Participants receive a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 165 mg/mL subcutaneously (SC); Cycle 2 Day 1: pembrolizumab 200 mg intravenously (IV); Cycle 3 Day 1: pembrolizumab 130 mg/mL SC; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
  Interventions: Biological: Pembrolizumab Dose C; Biological: Pembrolizumab Dose A; Biological: Pembrolizumab Dose B
- Cohort A Pembrolizumab Treatment Sequence 2 (Experimental): Participants receive a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 165 mg/mL SC; Cycle 2 Day 1: pembrolizumab 130 mg/mL SC; Cycle 3 Day 1: pembrolizumab 200 mg IV; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
  Interventions: Biological: Pembrolizumab Dose C; Biological: Pembrolizumab Dose A; Biological: Pembrolizumab Dose B
- Cohort A Pembrolizumab Treatment Sequence 3 (Experimental): Participants receive a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 130 mg/mL SC; Cycle 2 Day 1: pembrolizumab 165 mg/mL SC; Cycle 3 Day 1: pembrolizumab 200 mg IV; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
  Interventions: Biological: Pembrolizumab Dose C; Biological: Pembrolizumab Dose A; Biological: Pembrolizumab Dose B
- Cohort A Pembrolizumab Treatment Sequence 4 (Experimental): Participants receive a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 200 mg SC; Cycle 2 Day 1: pembrolizumab 200 mg IV; Cycle 3 Day 1: pembrolizumab 130 mg/mL SC; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab Dose 200 mg IV.
  Interventions: Biological: Pembrolizumab Dose C; Biological: Pembrolizumab Dose A; Biological: Pembrolizumab Dose B
- Cohort A Pembrolizumab Treatment Sequence 5 (Experimental): Participants receive a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 200 mg IV; Cycle 2 Day 1: pembrolizumab 130 mg/mL SC; Cycle 3 Day 1: pembrolizumab 165 mg/mL SC: Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
  Interventions: Biological: Pembrolizumab Dose C; Biological: Pembrolizumab Dose A; Biological: Pembrolizumab Dose B
- Cohort A Pembrolizumab Treatment Sequence 6 (Experimental): Participants receive a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 200 mg IV; Cycle 2 Day 1: pembrolizumab 165 mg/mL SC; Cycle 3 Day 1: pembrolizumab 130 mg/mL SC; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
  Interventions: Biological: Pembrolizumab Dose C; Biological: Pembrolizumab Dose A; Biological: Pembrolizumab Dose B
- Cohort B Pembrolizumab 400 mg IV (Experimental): Participants receive a single dose of pembrolizumab 400 mg IV on Day 1 of each 42-day cycle (every 6 weeks; Q6W) for up to 18 cycles (up to approximately 2 years).
  Interventions: Biological: Pembrolizumab Dose D

INTERVENTIONS:
Biological: Pembrolizumab Dose C — 165 mg/mL administered to a final dose of 285 mg via subcutaneous injection
  Other Names: KEYTRUDA®, MK-3475
  Arms: Cohort A Pembrolizumab Treatment Sequence 1; Cohort A Pembrolizumab Treatment Sequence 2; Cohort A Pembrolizumab Treatment Sequence 3; Cohort A Pembrolizumab Treatment Sequence 4; Cohort A Pembrolizumab Treatment Sequence 5; Cohort A Pembrolizumab Treatment Sequence 6
Biological: Pembrolizumab Dose A — 130 mg/mL administered to a final dose of 285 mg via subcutaneous injection
  Other Names: KEYTRUDA®, MK-3475
  Arms: Cohort A Pembrolizumab Treatment Sequence 1; Cohort A Pembrolizumab Treatment Sequence 2; Cohort A Pembrolizumab Treatment Sequence 3; Cohort A Pembrolizumab Treatment Sequence 4; Cohort A Pembrolizumab Treatment Sequence 5; Cohort A Pembrolizumab Treatment Sequence 6
Biological: Pembrolizumab Dose B — 200 mg administered via intravenous infusion
  Other Names: KEYTRUDA®, MK-3475
  Arms: Cohort A Pembrolizumab Treatment Sequence 1; Cohort A Pembrolizumab Treatment Sequence 2; Cohort A Pembrolizumab Treatment Sequence 3; Cohort A Pembrolizumab Treatment Sequence 4; Cohort A Pembrolizumab Treatment Sequence 5; Cohort A Pembrolizumab Treatment Sequence 6
Biological: Pembrolizumab Dose D — 400 mg administered via intravenous infusion
  Other Names: KEYTRUDA®, MK-3475
  Arms: Cohort B Pembrolizumab 400 mg IV

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic (PK) profile of pembrolizumab (MK-3475) following single subcutaneous (SC) injection of pembrolizumab Dose A versus pembrolizumab Dose C in adults with advanced melanoma. Additionally, the safety and tolerability of pembrolizumab SC injections will be assessed. And, finally, the efficacy of pembrolizumab intravenous (IV) infusion administration will be assessed.

DETAILED DESCRIPTION:
This study consists of two cohorts. Participants in Cohort A are randomized to one of six treatment sequences which will include 2 cycles of pembrolizumab administered via subcutaneous injection and 1 cycle of intravenous (IV) infusion, followed by up to 32 cycles (up to ~2 years) of pembrolizumab administered via IV infusion (each cycle is 21 days). Participants in Cohort B will receive pembrolizumab via IV infusion on Day 1 of each 21-day cycle for up to 18 cycles, up to ~ 2 years. Each cycle is 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of advanced melanoma.
* Has unresectable Stage III or Stage IV melanoma, as per American Joint Committee on Cancer (AJCC) staging system not amenable to local therapy.
* Has been untreated for advanced or metastatic disease except as follows:
* a. BRAF V600 mutant melanoma may have received standard of care targeted therapy (e.g. BRAF/ mitogen-activated protein kinase kinase enzyme [MEK] inhibitor, alone or in combination) and be eligible for this study.
* b. Prior adjuvant (post-surgery) or neoadjuvant (pre-surgery) melanoma therapy is permitted if it was completed ≥4 weeks before randomization and all related AEs have either returned to baseline or stabilized (resolution of toxic effect[s] of the most recent prior therapy to Grade 1 or less [except alopecia]).
* Female participants must agree to use contraception during the treatment period and for ≥120 days after the last dose of study treatment.
* Has measurable disease per RECIST 1.1 as assessed by BICR. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has adequate organ function.

Exclusion Criteria:

* Has received prior systemic treatment for unresectable or metastatic melanoma (exceptions as noted above in the Inclusion Criteria).
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. OX-40 and CD137) or any other antibody or drug specifically targeting checkpoint pathways other than anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) which is permitted in the adjuvant setting.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has ocular melanoma.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (15):
- Australia (6):
  - Orange Health Services ( Site 0004), Orange, New South Wales
  - Calvary Mater Newcastle ( Site 0006), Waratah, New South Wales
  - Cairns and Hinterland Hospital and Health Service ( Site 0001), Cairns, Queensland
  - Royal Adelaide Hospital ( Site 0002), Adelaide, South Australia
  - Ballarat Health Services ( Site 0003), Ballarat
  - MNCCI Port Macquarie Base Hospital ( Site 0005), Port Macquarie
- South Africa (5):
  - MPOC ( Site 0027), Groenkloof Pretoria, Gauteng
  - WITS Clinical Research CMJAH Clinical Trial Site ( Site 0030), Johannesburg, Gauteng
  - The Medical Oncology Centre of Rosebank ( Site 0026), Johannesburg, Gauteng
  - Cape Town Oncology Trials Pty Ltd ( Site 0028), Kraaifontein, Western Cape
  - Sandton Oncology Medical Group PTY LTD ( Site 0029), Johannesburg
- Spain (3):
  - Hospital Universitari Vall d Hebron ( Site 0062), Barcelona
  - Hospital Clinic i Provincial de Barcelona ( Site 0061), Barcelona
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 0063), Donostia / San Sebastian
- Karolinska Universitetssjukhuset Solna ( Site 0040), Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cohen G, Rapoport B, Chan SW, Ruff P, Arance A, Mujika Eizmendi K, Houghton B, Brown MP, Zielinski RM, Munoz Couselo E, Lyle M, Anderson JR, Jain L, de Alwis D, Lala M, Akala O, Chartash E, Jacobs C. Pembrolizumab 400 mg every 6 weeks as first-line therapy for advanced melanoma (KEYNOTE-555): Results from cohort B of an open-label, phase 1 study. PLoS One. 2024 Nov 12;19(11):e0309778. doi: 10.1371/journal.pone.0309778. eCollection 2024. PMID 39531423
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 138 participants were randomized and 137 participants received at least one dose of study intervention.
Groups:
- Cohort A Pembrolizumab Treatment Sequence 1: Participants received a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 165 mg/mL subcutaneously (SC); Cycle 2 Day 1: pembrolizumab 200 mg intravenously (IV); Cycle 3 Day 1: pembrolizumab 130 mg/mL SC; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
- Cohort A Pembrolizumab Treatment Sequence 2: Participants received a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 165 mg/mL SC; Cycle 2 Day 1: pembrolizumab 130 mg/mL SC; Cycle 3 Day 1: pembrolizumab 200 mg IV; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
- Cohort A Pembrolizumab Treatment Sequence 3: Participants received a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 130 mg/mL SC; Cycle 2 Day 1: pembrolizumab 165 mg/mL SC; Cycle 3 Day 1: pembrolizumab 200 mg IV; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
- Cohort A Pembrolizumab Treatment Sequence 4: Participants received a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 200 mg SC; Cycle 2 Day 1: pembrolizumab 200 mg IV; Cycle 3 Day 1: pembrolizumab 130 mg/mL SC; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab Dose 200 mg IV.
- Cohort A Pembrolizumab Treatment Sequence 5: Participants received a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 200 mg IV; Cycle 2 Day 1: pembrolizumab 130 mg/mL SC; Cycle 3 Day 1: pembrolizumab 165 mg/mL SC: Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
- Cohort A Pembrolizumab Treatment Sequence 6: Participants received a single dose of pembrolizumab in each 21-day cycle in the following sequence: Cycle 1 Day 1: pembrolizumab 200 mg IV; Cycle 2 Day 1: pembrolizumab 165 mg/mL SC; Cycle 3 Day 1: pembrolizumab 130 mg/mL SC; Cycle 4 Day 1 and every cycle thereafter, up to a total of 35 cycles (up to approximately 2 years), Day 1: pembrolizumab 200 mg IV.
- Cohort B Pembrolizumab 400 mg IV: Participants received a single dose of pembrolizumab 400 mg IV on Day 1 of each 42-day cycle (every 6 weeks; Q6W) for up to 18 cycles (up to approximately 2 years).
Period: Period 1
Arm/Group | Cohort A Pembrolizumab Treatment Sequence 1 | Cohort A Pembrolizumab Treatment Sequence 2 | Cohort A Pembrolizumab Treatment Sequence 3 | Cohort A Pembrolizumab Treatment Sequence 4 | Cohort A Pembrolizumab Treatment Sequence 5 | Cohort A Pembrolizumab Treatment Sequence 6 | Cohort B Pembrolizumab 400 mg IV
Started | 7 | 6 | 6 | 6 | 5 | 7 | 101
Treated | 7 | 6 | 6 | 5 | 5 | 7 | 101
Completed | 6 | 6 | 6 | 4 | 5 | 7 | 51
Not Completed | 1 | 0 | 0 | 2 | 0 | 0 | 50
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 45
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 5
Period: Period 2
Arm/Group | Cohort A Pembrolizumab Treatment Sequence 1 | Cohort A Pembrolizumab Treatment Sequence 2 | Cohort A Pembrolizumab Treatment Sequence 3 | Cohort A Pembrolizumab Treatment Sequence 4 | Cohort A Pembrolizumab Treatment Sequence 5 | Cohort A Pembrolizumab Treatment Sequence 6 | Cohort B Pembrolizumab 400 mg IV
Started | 6 | 6 | 6 | 4 | 5 | 7 | 0
Treated | 6 | 6 | 6 | 4 | 4 | 7 | 0
Completed | 6 | 6 | 6 | 4 | 5 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Cohort A Pembrolizumab Treatment Sequence 1 | Cohort A Pembrolizumab Treatment Sequence 2 | Cohort A Pembrolizumab Treatment Sequence 3 | Cohort A Pembrolizumab Treatment Sequence 4 | Cohort A Pembrolizumab Treatment Sequence 5 | Cohort A Pembrolizumab Treatment Sequence 6 | Cohort B Pembrolizumab 400 mg IV
Started | 6 | 6 | 6 | 4 | 5 | 6 | 0
Treated | 6 | 6 | 6 | 4 | 4 | 6 | 0
Completed | 6 | 5 | 6 | 4 | 4 | 6 | 0
Not Completed | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 4
Arm/Group | Cohort A Pembrolizumab Treatment Sequence 1 | Cohort A Pembrolizumab Treatment Sequence 2 | Cohort A Pembrolizumab Treatment Sequence 3 | Cohort A Pembrolizumab Treatment Sequence 4 | Cohort A Pembrolizumab Treatment Sequence 5 | Cohort A Pembrolizumab Treatment Sequence 6 | Cohort B Pembrolizumab 400 mg IV
Started | 6 | 5 | 6 | 4 | 4 | 6 | 0
Treated | 6 | 5 | 6 | 4 | 3 | 6 | 0
Completed | 3 | 1 | 2 | 2 | 3 | 6 | 0
Not Completed | 3 | 4 | 4 | 2 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 2 | 2 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Pembrolizumab Treatment Sequence 1 | Cohort A Pembrolizumab Treatment Sequence 2 | Cohort A Pembrolizumab Treatment Sequence 3 | Cohort A Pembrolizumab Treatment Sequence 4 | Cohort A Pembrolizumab Treatment Sequence 5 | Cohort A Pembrolizumab Treatment Sequence 6 | Cohort B Pembrolizumab 400 mg IV | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 5 | 7 | 101 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (14.9) | 54.0 (20.1) | 58.2 (12.4) | 49.8 (16.7) | 59.8 (18.0) | 63.0 (22.5) | 62.1 (13.9) | 60.9 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3 | 1 | 2 | 36 | 45
  Male | 6 | 5 | 5 | 3 | 4 | 5 | 65 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 6 | 4 | 3 | 5 | 93 | 120
  Unknown or Not Reported | 2 | 2 | 0 | 2 | 2 | 2 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  White | 7 | 6 | 6 | 6 | 5 | 7 | 87 | 124
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve (AUC) of Pembrolizumab - Cohort A
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected at designated time points and a pharmacokinetic (PK) model based on historical intravenous pembrolizumab PK data were used for the determination of the AUC of pembrolizumab. Geometric least-square mean (GM) and 95% confidence intervals were derived from mixed-effects model performed on natural log-transformed values. Data were reported by treatment received.
Time Frame: Cycles 1-3: Day 1 Predose and Days 2, 5, 10 and 15; Cycle 4: Day 1 Predose. Samples were also collected after IV infusion on Cycles 1-3: Day 1 ~0.5 hours after infusion and after SC injection on Days 3, 4, 6, and 7. Each cycle was 21 days.
Population: All participants in Cohort A who were complaint with the study procedures and had available data from IV treatment and at least one SC treatment cycle were analyzed per protocol by treatment. Per protocol, participants in Cohort B were analyzed separately.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg*day/L
Groups:
- Cohort A Pembrolizumab 130 mg/mL SC: Participants received pembrolizumab 130 mg/mL via subcutaneous injection on Day 1 of a 21-day cycle.
- Cohort A Pembrolizumab 165 mg/mL SC: Participants received pembrolizumab 165 mg/mL via subcutaneous injection on Day 1 of a 21-day cycle.
- Cohort A Pembrolizumab 200 mg IV: Participants received pembrolizumab 200 mg via intravenous injection on Day 1 of a 21-day cycle.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV
Number analyzed (Participants) | 32 | 32 | 32
mg*day/L | 507 [440 to 585] | 480 [418 to 551] | 695 [631 to 766]
Statistical Analysis 1: Comparison: Cohort A Pembrolizumab 130 mg/mL SC vs Cohort A Pembrolizumab 200 mg IV; Test type: Other — Geometric Least-Square Mean Ratio (GMR) = GM of Pembrolizumab 130 mg/mL SC/GM of Pembrolizumab 200 mg IV; GMR = 0.73, 90% CI 2-sided [0.68 to 0.78]
Statistical Analysis 2: Comparison: Cohort A Pembrolizumab 165 mg/mL SC vs Cohort A Pembrolizumab 200 mg IV; Test type: Other — GMR = GM of Pembrolizumab 165 mg/mL SC/GM of Pembrolizumab 200 mg IV; GMR = 0.69, 90% CI 2-sided [0.64 to 0.74]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Pembrolizumab - Cohort A
Description: Cmax was defined as the maximum concentration of pembrolizumab observed in plasma following a single dose. Blood samples were collected at designated time points and a PK model based on historical intravenous pembrolizumab PK data were used for the determination of the AUC of pembrolizumab. GM and 95% confidence intervals were derived from mixed-effects model performed on natural log-transformed values. Data were reported by treatment received.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV
Number analyzed (Participants) | 32 | 32 | 32
mg/L | 28.6 [24.7 to 33.1] | 26.8 [23.2 to 30.9] | 71.3 [65.6 to 77.5]
Statistical Analysis 1: Comparison: Cohort A Pembrolizumab 130 mg/mL SC vs Cohort A Pembrolizumab 200 mg IV; Test type: Other — GMR = GM of Pembrolizumab 130 mg/mL SC/GM of Pembrolizumab 200 mg IV; Geometric Least-Square Mean Ratio = 0.40, 90% CI 2-sided [0.36 to 0.44]
Statistical Analysis 2: Comparison: Cohort A Pembrolizumab 165 mg/mL SC vs Cohort A Pembrolizumab 200 mg IV; Test type: Other — GMR = GM of Pembrolizumab 165 mg/mL SC/GM of Pembrolizumab 200 mg IV; Geometric Least-Square Mean Ratio = 0.38, 90% CI 2-sided [0.34 to 0.41]

3. Primary Outcome: Bioavailability (F) of Pembrolizumab - Cohort A
Description: Blood samples were collected at designated time points and a population PK model based on historical intravenous pembrolizumab PK data was used for the determination of the F of pembrolizumab. Per protocol, an integrated population PK analysis was performed and combined data for Cohort A was reported.
Time Frame: as for outcome 1
Population: All participants in Cohort A who were compliant with the study procedure and had available data from IV treatment and at least one SC treatment cycle were analyzed. Per protocol, data were pre-specified to be combined for participants in Cohort A; therefore data by individual dose were not analyzed. Participants in Cohort B weren't analyzed, per protocol.
Measure: Mean (95% Confidence Interval); unit: Percent
Groups:
- Combined Cohort A: On Day 1 of Cycle 1 through Cycle 4, participants received one dose of the following: pembrolizumab 130 mg/mL via subcutaneous injection, pembrolizumab 165 mg/mL via subcutaneous injection, or pembrolizumab 200 mg via intravenous injection, depending on randomized treatment sequence. Each cycle was 21 days.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV | Combined Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 32
Percent |  |  |  | 66 [58 to 74]

4. Primary Outcome: Absorption Rate Constant (Ka) of Pembrolizumab - Cohort A
Description: Blood samples were collected at designated time points and a population PK model based on historical intravenous pembrolizumab PK data was used for the determination of the Ka of pembrolizumab. Per protocol, an integrated population PK analysis was performed and combined data for Cohort A was reported. Participants in Cohort B weren't analyzed, per protocol.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Error); unit: 1/day
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV | Combined Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 32
1/day |  |  |  | 0.191 (13.1)

5. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Pembrolizumab - Cohort A
Description: Blood samples were collected at designated time points for the determination of the Tmax of pembrolizumab.
Time Frame: as for outcome 1
Population: All participants in Cohort A who were complaint with the study procedures and had available data from IV treatment and at least one SC treatment cycle were analyzed per protocol by treatment. Per protocol, participants in Cohort B were not analyzed.
Measure: Median (Full Range); unit: Days
Groups:
- Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3): Participants received pembrolizumab 200 mg via intravenous injection on Day 1 of a 21-day cycle.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3)
Number analyzed (Participants) | 32 | 32 | 32
Days | 6.55 [3.70 to 21.00] | 8.35 [3.00 to 21.00] | 0.02 [0.02 to 0.02]

6. Primary Outcome: Clearance (CL) of Pembrolizumab - Cohort A
Description: Blood samples were collected at designated time points and a population PK model based on historical intravenous pembrolizumab PK data was used for the determination of the CL of pembrolizumab. Per protocol, an integrated population PK analysis was performed and combined data for Cohort A was reported.
Time Frame: as for outcome 1
Population: All participants who were complaint with the study procedures and had available data from IV treatment and at least one SC treatment cycle were analyzed. Per protocol, data were pre-specified to be combined for participants in Cohort A; therefore data by individual dose were not analyzed. Participants in Cohort B weren't analyzed, per protocol.
Measure: Mean (Standard Error); unit: Liters/day
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV | Combined Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 32
Liters/day |  |  |  | 0.25 (6.28)

7. Primary Outcome: Central Volume of Distribution (Vc) of Pembrolizumab - Cohort A
Description: Blood samples were collected at designated time points and a population PK model based on historical intravenous pembrolizumab PK data was used for the determination of the Vc of pembrolizumab. Per protocol, an integrated population PK analysis was performed and combined data for Cohort A was reported.
Time Frame: as for outcome 1
Population: All participants in Cohort A who were complaint with the study procedures and had available data from IV treatment and at least one SC treatment cycle were analyzed. Per protocol, data were pre-specified to be combined for participants in Cohort A; therefore data by individual dose were not analyzed. Participants in Cohort B weren't analyzed, per protocol.
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV | Combined Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 32
Liters |  |  |  | 3.39 (5.68)

8. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Cohort B
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions). Responses were based upon blinded independent central review (BICR) per RECIST 1.1. ORR was reported for participants in Cohort B.
Time Frame: Up to approximately 54 months
Population: All randomized participants in Cohort B who received at least one dose of study intervention were analyzed. Per protocol, participants in Cohort A were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 101
Percentage of Participants | 53.5 [43.3 to 63.5]

9. Secondary Outcome: Number of Participants Positive for Pembrolizumab Anti-Drug Antibody (ADA) Formation - Cohort A
Description: Blood samples were collected at designated time points for the determination of the presence or absence of pembrolizumab anti-drug antibodies. The number of participants who develop anti-pembrolizumab antibodies were assessed in Cycles 1 through Cycle 4. Per ADA immunogenicity analysis report, data from participants in Cohort A were reported combined across treatment cycles 1-4.
Time Frame: Cycles 1-4 Day 1: Predose. Each cycle is 21 days. (Up to approximately 64 days)
Population: All randomized participants in Cohort A who had at least one, conclusive ADA sample available after treatment with pembrolizumab in Cycles 1 through Cycle 4 were analyzed. Participants in Cohort B weren't analyzed, per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Pembrolizumab 130 mg/mL SC: Participants received pembrolizumab 130 mg/mL via subcutaneous injection on Day 1 of a 21 day cycle.
- Cohort A Pembrolizumab 165 mg/mL SC: Participants received pembrolizumab 165 mg/mL via subcutaneous injection on Day 1 of a 21 day cycle.
- Cohort A Pembrolizumab 200 mg IV: Participants received pembrolizumab 200 mg via intravenous injection on Day 1 of a 21 day cycle.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV | Combined Cohort A
Number analyzed (Participants) | 0 | 0 | 0 | 25
Participants |  |  |  | 0

10. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Event (AEs) - Cohort A
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced one or more AEs in Cohort A was reported. Per protocol, data were reported by treatment received and AEs from Cycles 4-35 were reported separately.
Time Frame: Up to approximately 27 months
Population: All randomized participants in Cohort A who received at least one dose of study intervention were analyzed. Per protocol, AEs from Cycles 4-35 were reported separately and participants in Cohort B were analyzed separately.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Pembrolizumab 165 mg/mL SC: Participants received pembrolizumab 130 mg/mL via subcutaneous injection on Day 1 of a 21-day cycle.
- Cohort A Pembrolizumab 200 mg IV (Cycle 4 - Cycle 35): In Cycle 4 through Cycle 35, participants received pembrolizumab 200 mg via intravenous injection on Day 1 of each 21-day cycle.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3) | Cohort A Pembrolizumab 200 mg IV (Cycle 4 - Cycle 35)
Number analyzed (Participants) | 33 | 34 | 34 | 30
Participants | 18 | 18 | 14 | 29

11. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE - Cohort A
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued due to an AE in Cohort A were reported. Per protocol, data were reported by treatment received and data from Cycles 4-35 were reported separately.
Time Frame: Up to approximately 23 months
Population: All participants in Cohort A who received at least one dose of study intervention were analyzed. All randomized participants in Cohort A who received at least one dose of study intervention were analyzed. Per protocol, data from Cycles 4-35 were reported separately and participants in Cohort B were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3) | Cohort A Pembrolizumab 200 mg IV (Cycle 4 - Cycle 35)
Number analyzed (Participants) | 33 | 34 | 34 | 30
Participants | 1 | 0 | 1 | 5

12. Secondary Outcome: Number of Participants With One or More Injection Site Signs and Symptoms After Subcutaneous Pembrolizumab Injection in Cycles 1-3 - Cohort A
Description: Participants completed the Injection Site Signs and Symptoms Questionnaire, within 60 minutes after each pembrolizumab SC injection during Cycles 1-3. Participants rated any pain, itching, swelling and redness they experienced at the pembrolizumab SC injection site from "None" to "Severe". The number of participants who experienced an injection site sign or symptom was reported.
Time Frame: Cycles 1-3 Day 1: Up to 60 minutes postdose. Each cycle is 21 days. (Up to approximately 43 days)
Population: Per protocol, participants in Cohort A who received a subcutaneous dose of pembrolizumab were analyzed by treatment received. Therefore, data were not analyzed in participants who received IV infusion. Participants in Cohort B were not analyzed, per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3): Participants received pembrolizumab 200 mg via intravenous injection on Day 1 of a 21 day cycle.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3)
Number analyzed (Participants) | 33 | 34 | 0
Participants | 3 | 2 |

13. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 - Cohort B
Description: For participants who demonstrated a CR (disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR was calculated for RECIST 1.1 based on BICR. DOR for Cohort B was reported.
Time Frame: Up to approximately 54 months
Population: All randomized participants in Cohort B who received at least one dose of study intervention and demonstrated a confirmed CR or PR response were analyzed. Per protocol, participants in Cohort A were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 54
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of responding participants with relapse.

14. Secondary Outcome: Progression-free Survival (PFS) Per to RECIST v1.1 Modified to Follow a Maximum of 10 Target Lesions and a Maximum of 5 Target Lesions Per Organ - Cohort B
Description: PFS was defined as the time from the first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Although RECIST 1.1 was modified to allow for a maximum of 10 target lesions in total and 5 per organ. Per protocol, PFS as assessed by BICR for participants in Cohort B was reported.
Time Frame: Up to approximately 54 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 101
Months | 13.8 [5.3 to 41.4]

15. Secondary Outcome: Overall Survival (OS) - Cohort B
Description: OS was defined as the time from the first dose of study treatment to death due to any cause. Per protocol, OS for participants in Cohort B was reported.
Time Frame: Up to approximately 54 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 101
Months | NA [27.1 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

16. Secondary Outcome: Early Cycle AUC of Pembrolizumab - Cohort B
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected at designated time points for the determination of the pembrolizumab AUC in participants in Cohort B during Cycle 1 (early cycle). Blood samples were also collected predose on Day 1 of Cycle 2 just prior to the next dose as the last sample (trough concentration) of Cycle 1. A cycle was 42 days.
Time Frame: Cycle 1: Day 1 Predose and ~5 minutes post infusion and Day 22; Cycle 2: Predose. A Cycle was 42 days. (Up to approximately 6 weeks)
Population: All randomized participants in Cohort B who were compliant with the study procedures and had available data at the specified time point were analyzed. Per protocol, participants in Cohort A were analyzed separately.
Measure: Median (90% Confidence Interval); unit: μg/ml
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 101
μg/ml | NA [NA to NA] — AUC was determined by trapezoidal methods using interpolation between data points. Thus, at least 3 data points in the terminal phase excluding Tmax (i.e., end of infusion) were required to determine AUC. Due to sparse PK sampling schedule, per participant data could not be calculated.

17. Secondary Outcome: Steady State AUC of Pembrolizumab - Cohort B
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected at designated time points for the determination of the pembrolizumab AUC in participants in Cohort B during Cycle 4 (steady state). Blood samples were also collected predose on Day 1 of Cycle 5 just prior to the next dose as the last samples (trough concentration) of Cycle 4. Each cycle was 42 days.
Time Frame: Cycle 4: Day 1 Predose and ~5 minutes post infusion and Day 22; Cycle 5: Predose. A Cycle was 42 days. (Up to approximately 6 weeks)
Population: as for outcome 16
Measure: Median (90% Confidence Interval); unit: μg/ml
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 73
μg/ml | NA [NA to NA] — AUC was determined by trapezoidal methods using interpolation between data points. Thus, at least 3 data points in the terminal phase excluding Tmax (i.e., end of infusion) were required to determine AUC. Due to sparse PK sampling schedule, per participant data could not be calculated.

18. Secondary Outcome: Early Cycle Cmax of Pembrolizumab - Cohort B
Description: Cmax was defined as the maximum concentration of pembrolizumab observed in plasma following a single dose. Blood samples were collected at designated time points for the determination of the pembrolizumab Cmax in participants in Cohort B during Cycle 1 (early cycle). Blood samples were also collected predose on Day 1 of Cycle 2 just prior to the next dose as the last sample (trough concentration) of Cycle 1. Each cycle was 42 days.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Median (90% Confidence Interval); unit: μg/ml
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 99
μg/ml | 127.0 [121.3 to 132.7]

19. Secondary Outcome: Steady State Cmax of Pembrolizumab - Cohort B
Description: Cmax was defined as the maximum concentration of pembrolizumab observed in plasma following a single dose. Blood samples were collected at designated time points for the determination of the pembrolizumab Cmax in participants in Cohort B during Cycle 4 (steady state). Blood samples were also collected predose on Day 1 of Cycle 5 just prior to the next dose as the last sample (trough concentration) of Cycle 4. Each cycle was 42 days.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Median (90% Confidence Interval); unit: μg/ml
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 72
μg/ml | 150.0 [141.9 to 158.3]

20. Secondary Outcome: Early Cycle Minimum Plasma Concentration (Cmin) of Pembrolizumab - Cohort B
Description: Cmin was defined as the minimum concentration of pembrolizumab observed in plasma following a single dose. Blood samples were collected at designated time points for the determination of the pembrolizumab Cmin in participants in Cohort B during Cycle 1 (early cycle). Blood samples were also collected predose on Day 1 of Cycle 2 just prior to the next dose as the last sample (trough concentration) of Cycle 1. Each cycle was 42 days.
Time Frame: as for outcome 16
Population: All randomized participants in Cohort B who were compliant with the study procedures and had available data at the specified time point were analyzed. Per protocol, participants in Cohort A were not analyzed.
Measure: Median (90% Confidence Interval); unit: μg/ml
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 87
μg/ml | 15.1 [13.5 to 16.9]

21. Secondary Outcome: Steady State Cmin of Pembrolizumab - Cohort B
Description: Cmin was defined as the minimum concentration of pembrolizumab observed in plasma following a single dose. Blood samples were collected at designated time points for the determination of the pembrolizumab Cmin in participants in Cohort B during Cycle 4 (steady state). Blood samples were also collected predose on Day 1 of Cycle 5 just prior to the next dose as the last sample (trough concentration) of Cycle 4. Each cycle was 42 days.
Time Frame: Cycle 4: Day 1 Predose and ~5 minutes post infusion and Day 22; Cycle 5: Predose. Each Cycle was 42 days. (Up to approximately 6 weeks)
Population: as for outcome 20
Measure: Median (90% Confidence Interval); unit: μg/ml
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 69
μg/ml | 24.0 [20.6 to 27.9]

22. Secondary Outcome: Number of Participants Who Experienced One or More AEs - Cohort B
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced one or more AEs in Cohort B was reported.
Time Frame: Up to approximately 54 months
Population: All randomized participants in Cohort B who received at least one dose of study intervention were analyzed. Per protocol, participants in Cohort A were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 101
Participants | 101

23. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE - Cohort B
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued due to an AE in Cohort B were reported.
Time Frame: Up to approximately 26 months
Population: All randomized participants in Cohort B who received at least one dose of study intervention. Per protocol, participants in Cohort A were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Pembrolizumab 400 mg IV
Number analyzed (Participants) | 101
Participants | 8

ADVERSE EVENTS:
Time Frame: Up to approximately 54 months
Description: Serious and Other adverse events (AEs) includes all participants who received ≥1 dose of study drug. All-Cause Mortality includes all randomized participants. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Per protocol, data are reported by treatment received & data for Cohort A Cycles 4-35 was reported separately.
Arm/Group | Cohort A Pembrolizumab 130 mg/mL SC | Cohort A Pembrolizumab 165 mg/mL SC | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3) | Cohort A Pembrolizumab 200 mg IV (Cycle 4 - Cycle 35) | Cohort B Pembrolizumab 400 mg IV
All-Cause Mortality (participants affected / at risk) | 1/34 | 3/35 | 1/35 | 4/31 | 45/101
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/34 | 2/34 | 9/30 | 31/101
Other Adverse Events (participants affected / at risk) | 15/33 | 15/34 | 8/34 | 27/30 | 93/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Pembrolizumab 130 mg/mL SC (N=33) | Cohort A Pembrolizumab 165 mg/mL SC (N=34) | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3) (N=34) | Cohort A Pembrolizumab 200 mg IV (Cycle 4 - Cycle 35) (N=30) | Cohort B Pembrolizumab 400 mg IV (N=101)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated adverse reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Pembrolizumab 130 mg/mL SC (N=33) | Cohort A Pembrolizumab 165 mg/mL SC (N=34) | Cohort A Pembrolizumab 200 mg IV (Cycle 1 - Cycle 3) (N=34) | Cohort A Pembrolizumab 200 mg IV (Cycle 4 - Cycle 35) (N=30) | Cohort B Pembrolizumab 400 mg IV (N=101)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 16 (33)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (8)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (8)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 7 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 6 (9)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 5 (7) | 20 (33)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (9)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 6 (7) | 17 (21)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 11 (13)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 29 (34)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 10 (10)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 4 (6) | 8 (11)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 8 (13) | 14 (26)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 13 (17)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 13 (18)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (3) | 6 (18)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (13)
Blood phosphorus increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 3 (3)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (9)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 6 (13)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (25)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (14)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 7 (9) | 32 (57)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 11 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 12 (14)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (7)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 9 (12)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (6)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (12)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 11 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 6 (7) | 20 (29)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 5 (10) | 22 (31)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 25 (25)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03665597/Prot_SAP_000.pdf